CLINICAL TRIAL: NCT03553147
Title: Evaluation of the SARC-F Score as a Screening Tool for Undernutrition in a Geriatric Population
Acronym: GERIASARC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CHU-390; 2017-A03050-53 (Other: 2017-A03050-53)
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Sarcopenia; Denutrition
Keywords: denutrition screening tool; SARC-F score; denutrition in geriatric population; sarc-f score associated with denutrition
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group/Cohort 1 (Experimental): all patient SARC-F score, handgrip test and impedancemetry
  Interventions: Other: SARC-F score, handgrip test and impedancemetry

INTERVENTIONS:
Other: SARC-F score, handgrip test and impedancemetry — Participation in the study will be offered to any patient admitted to the geriatric ward, those who meet the inclusion criteria and do not have exclusion criteria will have to complete the SARC-F questionnaire during their stay, and to do the handgrip test and impedancemetry performed by a third party. Biological data (albumin, pre-albumin and C-Reactive Protein) and anthropometric data will be collected and analyzed to determine if the patient is malnourished or not, and the results of SARC-F will be compared between these 2 groups.

SUMMARY:
To study the relationship between sarcopenia and undernutrition in adult patients over 70 years of age, and at the same time to define a threshold value for the predictive SARC-F score of undernutrition.

Hypothesis : the SARC-F score is correlated with malnutrition defined according to the following HAS criteria :

Moderate denutrition Severe denutrition

DETAILED DESCRIPTION:
The geriatric population is a population at risk, given the frequent and numerous comorbidities present. Undernutrition is one of these, which is frequently associated with sarcopenia, that is, a decrease in muscle strength. Its screening must be early to avoid complications (osteoporosis, fractures, infections ...) and given the cost it generates for society. However, the detection of undernutrition can sometimes be time-consuming and its criteria in default, such as in the presence of edema or obesity, for example. There is a score, the SARC-F, which allows to detect sarcopenia from a result greater than or equal to 4, but which does not allow direct detection of undernutrition.

The primary objective is to evaluate the SARC-F score as a screening tool for undernutrition in a geriatric population, secondary objectives being to find a threshold value at this score, and also to estimate a prevalence of undernutrition in this population.

It will be a cross-sectional exploratory study to evaluate a diagnostic tool, the SARC-F score, with comparison between cases and controls.

The study will be conducted in a single center, a geriatric short-stay service. Participation in the study will be offered to any patient admitted to the geriatric ward, those who meet the inclusion criteria and do not have exclusion criteria will have to complete the SARC-F questionnaire during their stay, and to do the handgrip test and impedancemetry performed by a third party. Biological data (albumin, pre-albumin and C-Reactive Protein) and anthropometric data will be collected and analyzed to determine if the patient is malnourished or not, and the results of SARC-F will be compared between these 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* 70 years and over
* living at home or in nursing homes in Puy-de-Dôme
* sent in short geriatric stay at the Grand Pré clinic by their general practioner, an emergency department or an EHPAD

Exclusion Criteria:

* refusal to participate in the study
* severe dementia preventing answering SARC-F questions
* no fluency in the French language
* patient with a pacemaker (contraindication of the use of impedancemetry)

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
score SARC-F | at day 1
  SARC-F score (dependent variable) defined by a questionnaire, completed by the patient during the stay at the clinic. This questionnaire includes 5 questions rated from 0 to 2 and is therefore 10 in total. It is admitted the presence of sarcopenia for a score greater than or equal to 4 according to the literature. However, there is currently no study defining a threshold for the diagnosis of undernutrition

SECONDARY OUTCOMES:
SARC-F to predict undernutrition | at day 1
  discriminant values of SARC-F to predict undernutrition in the study population, considered qualitatively or quantitatively
denutrition prevalence | at day 1
  overall prevalence of undernutrition in the study population

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas FARIGON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Cederholm T, Bosaeus I, Barazzoni R, Bauer J, Van Gossum A, Klek S, Muscaritoli M, Nyulasi I, Ockenga J, Schneider SM, de van der Schueren MA, Singer P. Diagnostic criteria for malnutrition - An ESPEN Consensus Statement. Clin Nutr. 2015 Jun;34(3):335-40. doi: 10.1016/j.clnu.2015.03.001. Epub 2015 Mar 9. PMID 25799486
- [Background] Delliere S, Cynober L. Is transthyretin a good marker of nutritional status? Clin Nutr. 2017 Apr;36(2):364-370. doi: 10.1016/j.clnu.2016.06.004. Epub 2016 Jun 20. PMID 27381508
- [Background] Zamboni M, Mazzali G, Fantin F, Rossi A, Di Francesco V. Sarcopenic obesity: a new category of obesity in the elderly. Nutr Metab Cardiovasc Dis. 2008 Jun;18(5):388-95. doi: 10.1016/j.numecd.2007.10.002. Epub 2008 Apr 18. PMID 18395429
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Beaudart C, Zaaria M, Pasleau F, Reginster JY, Bruyere O. Health Outcomes of Sarcopenia: A Systematic Review and Meta-Analysis. PLoS One. 2017 Jan 17;12(1):e0169548. doi: 10.1371/journal.pone.0169548. eCollection 2017. PMID 28095426
- [Background] Deren ME, Babu J, Cohen EM, Machan J, Born CT, Hayda R. Increased Mortality in Elderly Patients with Sarcopenia and Acetabular Fractures. J Bone Joint Surg Am. 2017 Feb 1;99(3):200-206. doi: 10.2106/JBJS.16.00734. PMID 28145950
- [Background] Ethgen O, Beaudart C, Buckinx F, Bruyere O, Reginster JY. The Future Prevalence of Sarcopenia in Europe: A Claim for Public Health Action. Calcif Tissue Int. 2017 Mar;100(3):229-234. doi: 10.1007/s00223-016-0220-9. Epub 2016 Dec 24. PMID 28012107
- [Background] Malmstrom TK, Miller DK, Simonsick EM, Ferrucci L, Morley JE. SARC-F: a symptom score to predict persons with sarcopenia at risk for poor functional outcomes. J Cachexia Sarcopenia Muscle. 2016 Mar;7(1):28-36. doi: 10.1002/jcsm.12048. Epub 2015 Jul 7. PMID 27066316
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716